CLINICAL TRIAL: NCT06203288
Title: Short-Term & Long-Term Benefits for Enhancing Educator & Student Prosocial Behavior, Well-being, & Resilience Through Mindfulness-Based Social and Emotional Learning Programs in Schools
Brief Title: Well-being in Students and Teachers Study
Acronym: WIST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY2023-1289
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Prosocial Behavior; Community Sense; Optimism; Anxiety; Social Competence; Self-Compassion; Stress, Psychological; Burnout, Professional; Efficacy, Self; Self Awareness
Keywords: social and emotional learning; SEL; mindfulness-based intervention; MBI
MeSH Terms: conditions — Altruism; Anxiety Disorders; Social Skills; Stress, Psychological; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MBSEL program for educators (Experimental): Teachers randomized to this arm will receive a mindfulness-based social and emotional learning (MBSEL) program for educators training outside the classroom. These teachers will continue to teach their regular "business as usual" social and emotional learning (SEL) curriculum in the classroom.
  Note: In the school district where this research study is being conducted, every teacher is required to allot at least one 50-min class period to implementing SEL programs and/or practices, and to embed SEL activities and practices throughout the school day.
  Interventions: Behavioral: Mindfulness-based social and emotional learning (MBSEL) program for educators
- MBSEL program for educators and MBSEL program for students (Experimental): Teachers randomized to this arm will first receive training in a mindfulness-based social and emotional learning (MBSEL) program designed specifically for educators and will complete the program on their own outside the classroom. Following, they will receive training for implementing an MBSEL program for their students, and then they implement weekly lessons of this program in their classroom to their students.
  Interventions: Behavioral: Mindfulness-based social and emotional learning (MBSEL) program for educators; Behavioral: Mindfulness-based social and emotional learning (MBSEL) program for students
- Comparison "Business as Usual" (No Intervention): Teachers randomized to this arm will teach their regular "business as usual" social and emotional learning (SEL) curriculum to their student in the classroom.
  Note: In the school district where this research study is being conducted, every teacher is required to allot at least one 50-min class period to implementing SEL programs and/or practices, and to embed SEL activities and practices throughout the school day.

INTERVENTIONS:
Behavioral: Mindfulness-based social and emotional learning (MBSEL) program for educators — MBSEL for educators is a program designed to improve teachers' ability to deal with stress and enhance their well-being and teaching. Lessons include: (1) Introduction to the Science, (2) Brain, Attention, & Well-being, (3) Positive Neuroscience, (4) Mindful Teaching, (5) Embracing Self-Compassion, (6) Finding Your Compass: Intentions for Mindful Living. This 2-hour program is self-paced and delivered online.
  Arms: MBSEL program for educators; MBSEL program for educators and MBSEL program for students
Behavioral: Mindfulness-based social and emotional learning (MBSEL) program for students — MBSEL program for students consists of 17 lessons taught about once a week (40-50 minutes per lesson). The core mindfulness program practices (done every day for 3 minutes three times a day) consist of focusing on one's breathing and attentive listening to a single resonant sound. The lessons focus on promoting prosocial behavior (e.g., kindness, altruism), resiliency, well-being, and reducing stress in students. It also incorporates an eco-behavioral systems orientation.
  Arms: MBSEL program for educators and MBSEL program for students

SUMMARY:
The goal of this randomized trial is to test the effectiveness of two universal classroom-based mindfulness social and emotional learning (SEL) programs (one for students and one for teachers) by examining behavioral outcomes on 5th and 6th grade students and their teachers. The main questions it aims to answer are:

* What are the singular and combined effects of a mindfulness-based SEL education programs for teachers and their students on the development of students' and their teachers' social, emotional, and cognitive competence, and well-being?
* Can mindfulness-based SEL education programs for students and teachers foster the creation of caring, inclusive, equitable, and collaborative classroom contexts?
* Can mindfulness-based SEL education programs support the development of students' and teachers' prosocial attitudes, mindsets that positively impact student learning?
* Are the effects durable beyond the end of the programs with regard to the singular and combined mindfulness-based SEL interventions?

A total of 24 classrooms will be randomized into one of three study conditions:

1. Mindfulness SEL program for Educators only
2. Mindfulness SEL program for Educators and Mindfulness SEL program for Students in combination, and
3. "Business as usual" (comparison groups in which regular classroom SEL curricula is implemented).

Data will be obtained via multiple objective and subjective methods (e.g., self- and teacher-reports, peer behavioral assessments) from different sources (e.g., self-, peer-, and teacher-reports). Data will also be collected to monitor implementation of the two programs. To explore the ways in which these two programs impact student, teacher, and classroom outcomes, data will be analyzed to compare students and teachers in the three conditions. In Phase One (year one), the investigators will conduct an experimental "outcome" study to examine the singular and combined effects of the two programs by comparing pre-test and post-test measures across the three conditions. In Phase Two (year two), the investigators will conduct a six-month follow up with those teachers and students who participated in Phase One in order to determine the degree to which the program effects are durable after the program has ended.

DETAILED DESCRIPTION:
Project Description: This research is designed to address a lacuna in the field by examining the effectiveness of two universal mindfulness-based social and emotional learning (MBSEL) classroom programs that focus on promoting social, emotional, and cognitive competence and positive classroom environments for early adolescent students and their teachers. Specifically, we will test the effectiveness of an MBSEL program for students and an MBSEL program for teachers, both singularly (MBSEL for teachers) and in combination (educator and students) and examine short-term and long-term outcomes on student and teacher behaviors. The study represents a critical advance in the field of education by exploring the short-term and long-term effects of two programs, singularly and in combination, and will be the first to explore student and teacher outcomes on multiple social, emotional, cognitive, motivational, behavioral, and classroom systems via multiple methods. The focus of the study is on early adolescence - a distinctive time period in which individuals undergo important developmental changes and critical developmental transitions occur.

Project Significance: The escalating mental health crisis in our children and youth has ignited a call to action for finding effective preventive programs that can deter mental health problems before they begin. Indeed, the crisis of children's mental health and rising disparities in educational outcomes has risen to the forefront of national consciousness with the release of the most recent U.S. Surgeon General's Advisory in December 2021. The Advisory calls attention to the rising mental health issues of young people and disparities across subpopulations in the U.S. It then outlines a whole-society approach for tackling the problem and includes a set of recommendations designed to prevent these challenges and bolster children's well-being. One of the primary recommendations outlined is to "support the mental health of children and youth in educational, community, and childcare settings," which involves, "creating positive, safe, and affirming educational environments" and "expanding programming that promotes healthy development (such as social and emotional learning)". To support the well-being and mental health of students, the Advisory also encourages policymakers and schools to undertake efforts designed to promote the "mental health of all school personnel". The Advisory proports that these efforts will directly benefit school personnel, while at the same time, help to foster teachers' social and emotional competencies (SECs), including empathy and compassion-competencies that are needed to create positive learning environments that can promote student well-being and healthy development. Furthermore, other policy makers and advocacy groups in the U.S. have called for the increased training of teachers in SEL so that teachers are better equipped to support the development of students' well-being.

The present study is novel in several ways. First, it represents an initial study to examine the effectiveness an MBSEL education program on a wide corpus of both teacher and student level outcomes. That is, it will examine if a program that is directed to cultivating teacher well-being and prosociality can have collateral benefits for students. Second, it is the first attempt to explore the "value - added" of integrating an MBSEL program for teachers with an already well-established and well-researched MBSEL program for students. Indeed, several studies have demonstrated the effectiveness of MBSEL programs on students' well-being, cognitive control, and prosocial behaviors, yet no research to date has examined the extent to which there are additional benefits to teachers and students if teachers also receive an MBSEL program for themselves before they implement a program for students. Third, the study will utilize a longitudinal design to examine the durability of the effects of the two programs, both singularly and jointly after the programs have ended.

The investigators see joint efforts geared towards supporting the well-being and social and emotional competencies of both teachers and students as an effective approach to address the rising trends in mental health challenges and to build optimal learning environments for students to develop, thrive and feel fully included. However, a paucity of research has explored how teachers impact the development of students' social and emotional competencies nor has it explored how teachers' own social and emotional competencies impact that of students. Furthermore, little research has tested the impacts of programming designed to develop teacher social and emotional competencies on student outcomes and/or whether these teachers are more capable of creating inclusive classroom environments that foster equitable educational outcomes. Failure to understand the role of teachers in cultivating students' social and emotional competencies and the lack of insight on how best to support teachers' own well-being and social and emotional competence has led to a gap in knowledge regarding whether and how best to promote students' social and emotional competencies and a classroom climate that supports the prosocial behavior, mental health and well-being of students.

Study Aims and Conceptual Framework The goal of this study is to evaluate the single and joint effects of a universal MBSEL program for early adolescent students, and a companion program for teachers on multiple individual and contextual outcomes and to examine both the short-term and long-term effects of these interventions. In conceptualizing and designing this study, the investigators draw from a developmental systems perspective that "recognizes that human development is a bi-directional, individual ↔ context relational process" in which "there are multiple levels of organization within the individual (e.g., motivation, and cognitive abilities) that influence one's development course," and "different levels of organization within the social ecology (e.g., families, schools, and neighborhoods) that contribute to development".

The investigators have identified the time of early adolescence to be a crucial time for promoting prosociality (e.g., empathy, compassion, kindness, altruism), curbing mental health issues, and altering students' personal and academic trajectories. Indeed, one period of development in which MBSEL programs may be particularly beneficial is during the transition to adolescence. The early adolescent years are a time of psychological and social change associated with the onset of many mental health problems and declines in well-being.

Findings from studies of mindfulness-based interventions (MBIs) with teachers indicate promising benefits for teachers and their classroom practices, however, less is known about the impact these trainings directly have on their students. Several studies show that teacher mindfulness programs are effective in reducing teacher stress and bolstering their well-being. Furthermore, a recent review of studies of MBIs with teachers found that, on average, MBIs generated improvements in mindfulness, well-being, job satisfaction, empathy, compassion, resilience, and emotion regulation, as well as reductions in stress, burnout, anxiety, and depression.

Therefore, more research is needed to explore the effects of mindfulness training for teachers on their ability to implement mindfulness programming with youth and the impact it has on student and classroom outcomes. That said, the investigators do know that teacher mindfulness is related to a host of positive outcomes for their own lives, their teaching, and for that of their students. Recent research has also found that student perceptions of their teachers' mindful qualities predict changes in their perceptions of school need fulfillment (i.e., the idea that their school meets their basic needs for autonomy, competence, and relatedness). These changes in turn predict changes in students' own mindfulness, self-compassion, and compassion for others over the course of the school year. In other words, how students perceive their teachers' mindful qualities impacts their own development.

In light of the initial findings from recent studies, research is needed on how best to develop the skills of mindfulness and other social and emotional competencies in teachers so that they are adequately prepared and well equipped to cultivate these capacities in their students. It is important to consider approaches that allow for flexibility and a reasonable demand of teachers' time given their increasingly busy and stressful workloads. That said, trainings must not sacrifice competency for brevity and ease. The investigators see this study as an opportunity to explore a novel, hybrid approach to training teachers in mindfulness and subsequently training them in the administration of a mindfulness-based SEL promotion program for their students.

Method Study Context The proposed study will take place in racially diverse schools in the Chicagoland area. Note that the investigators have received approval from a superintendent and administrators to conduct the study in a large school district in suburban Chicago.

Study Design and Participants This study will be carried out via a randomized controlled trial (RCT), pretest-post-test, control group (business as usual) longitudinal design. A total of 24 elementary school teachers and their 5th and 6th grade students will be invited to participate.

Interventions MBSEL Program for Students: Teachers randomly assigned to implement the MBSEL program to their students will attend a 1 day training session wherein they will be provided with the theoretical and empirical underpinnings of the program along with the program's goals. As a means of facilitating internal validity, all training will be conducted by one of the program developers. During the preintervention training, teachers will be provided with the curriculum manual in which lesson plans are explicitly delineated. The 1-day training session will include interactive discussions on SEL, the developmental characteristics of early adolescents' social and emotional competence, presentation of material through lecture, video and readings, and role-plays of curriculum instructional techniques.

MBSEL Program for Educators: Teacher training and fidelity. Teachers who are randomly assigned to the MBSEL program for Educators will participate in a one half-day program implementation. Teachers' participation will be elicited via weekly diaries and reflections on their experiences with the program.

Data Analysis Data will be analyzed via Hierarchical Linear Modeling (HLM) in which the unit of the analysis is at the level of randomization - the classroom. Moreover, data will be analyzed via analysis of covariance to analyze outcomes while controlling for various demographic variables (e.g., English as a Second Language status, gender, grade). A composite variable representing classroom implementation will be created to allow for an examination of interaction effects of program outcomes by level of program implementation (e.g., the degree to which the teacher implemented the various curriculum lessons). Qualitative data gathered via open-ended questions and interviews will be content analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 5th and 6th grade teachers (minimum .5 full time equivalent) and their students

Exclusion Criteria:

* Part-time teachers (less than .5 full time equivalent), substitute teachers, school counselors, school administrators, or other school staff

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Student Prosocial Behavior Scores measured with Peer Nominations at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Following the procedures outlined by Parkhurst and Asher (1992), unlimited and cross-gender peer nominations will be used to obtain independent assessments of prosociality, whereby students are asked to nominate (circle all the names of) classmates who fit particular behavioral characteristics: (1) share and cooperate, and (2) help other kids when they have a problem. This methodology is consistent with published investigations in which peers' ratings of behaviors are considered to be a reliable and valid way in which to assess students' social behaviors in a school context (Schonert-Reichl, 1999; Wentzel et al., 2004; Oberle et al., 2010). Students' nominations are standardized within each classroom, and a proportional nominations score is calculated per student for each of the behaviors. Higher scores indicate higher levels of prosocial behavior.
Mean Change from Baseline in Student Prosocial Behavior Scores measured with Peer Nominations at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Following the procedures outlined by Parkhurst and Asher (1992), unlimited and cross-gender peer nominations will be used to obtain independent assessments of prosociality, whereby students are asked to nominate (circle all the names of) classmates who fit particular behavioral characteristics: (1) share and cooperate, and (2) help other kids when they have a problem. This methodology is consistent with published investigations in which peers' ratings of behaviors are considered to be a reliable and valid way in which to assess students' social behaviors in a school context (Schonert-Reichl, 1999; Wentzel et al., 2004; Oberle et al., 2010). Students' nominations are standardized within each classroom, and a proportional nominations score is calculated per student for each of the behaviors. Higher scores indicate higher levels of prosocial behavior.
Mean Change from Baseline in Student Optimism Scores on the Optimism Subscale of the Resiliency Inventory at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Student self-report with a 9-item subscale (Noam & Goldstein, 1998; Song, 2003) measured on a 5-point Likert scale, where 1=Not at all like me, 2=A little bit like me, 3=Kind of like me, 4=A lot like me, 5=Always like me. Mean score calculated, with higher scores indicating higher levels of optimism. Five items are reverse scored.
Mean Change from Baseline in Student Optimism Scores on the Optimism Subscale of the Resiliency Inventory at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Student self-report with a 9-item subscale (Noam & Goldstein, 1998; Song, 2003) measured on a 5-point Likert scale, where 1=Not at all like me, 2=A little bit like me, 3=Kind of like me, 4=A lot like me, 5=Always like me. Mean score calculated, with higher scores indicating higher levels of optimism. Five items are reverse scored.
Mean Change from Baseline in Student Attention and Concentration Scores on the Attention and Concentration Subscale of the Teacher Social Competence Rating Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher-rating of students 7-item subscale (Kam & Greenberg, 1998) measured on a 6-point Likert scale, where 1=Almost Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Very Often, 6=Almost Always. Mean score calculated, with higher scores indicating higher levels of attention and concentration. Two items are reverse scored.
Mean Change from Baseline in Student Attention and Concentration Scores on the Attention and Concentration Subscale of the Teacher Social Competence Rating Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher-rating of students 7-item subscale (Kam & Greenberg, 1998) measured on a 6-point Likert scale, where 1=Almost Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Very Often, 6=Almost Always. Mean score calculated, with higher scores indicating higher levels of attention and concentration. Two items are reverse scored.
Mean Change from Baseline in Student Social and Emotional Competence Scores on the Social and Emotional Competence Subscale of the Teacher Social Competence Rating Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher-rating of students 7-item subscale (Kam & Greenberg, 1998) measured on a 6-point Likert scale, where 1=Almost Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Very Often, 6=Almost Always. Mean score calculated, with higher scores indicating higher levels of social and emotional competence. No reverse scored items.
Mean Change from Baseline in Student Social and Emotional Competence Scores on the Social and Emotional Competence Subscale of the Teacher Social Competence Rating Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher-rating of students 7-item subscale (Kam & Greenberg, 1998) measured on a 6-point Likert scale, where 1=Almost Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Very Often, 6=Almost Always. Mean score calculated, with higher scores indicating higher levels of social and emotional competence. No reverse scored items.
Mean Change from Baseline in Teacher Self-Compassion Scores on the Teacher Self-Compassion Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher self-report with a 9-item scale (Neff, 2003; Roeser et al., 2013) measured on a 5-point Likert scale, where 1=Not at all true of me, 2=Rarely True of me, 3=Somewhat true of me, 4=Often true of me, 5=Very true of me. Mean score calculated, with higher scores indicating higher levels of self-compassion. Three items are reverse scored.
Mean Change from Baseline in Teacher Self-Compassion Scores on the Teacher Self-Compassion Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher self-report with a 9-item scale (Neff, 2003; Roeser et al., 2013) measured on a 5-point Likert scale, where 1=Not at all true of me, 2=Rarely True of me, 3=Somewhat true of me, 4=Often true of me, 5=Very true of me. Mean score calculated, with higher scores indicating higher levels of self-compassion. Three items are reverse scored.
Mean Change from Baseline in Teacher Stress Scores on the Stress Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher self-report with a 7-item scale (Pettegrew & Wolf, 1982) measured on a 5-point Likert scale, where 1=Strongly Disagree, 2=Disagree, 3=Unsure, 4=Agree, 5=Strongly Agree. Mean score calculated, with higher scores indicating higher levels of stress. No reverse scored items.
Mean Change from Baseline in Teacher Stress Scores on the Stress Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher self-report with a 7-item scale (Pettegrew & Wolf, 1982) measured on a 5-point Likert scale, where 1=Strongly Disagree, 2=Disagree, 3=Unsure, 4=Agree, 5=Strongly Agree. Mean score calculated, with higher scores indicating higher levels of stress. No reverse scored items.
Mean Change from Baseline in Teacher Burnout Scores on the Maslach Burnout Inventory at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher self-report with a 23-item scale (Maslach & Jackson, 1981) measured on a 7-point Likert scale, where 1=Never, 2=A few times, 3=Once a month or less, 4=A few times a month, 5=Once a week, 6=A few times a week, 7=Every day. Mean score calculated, with higher scores indicating higher levels of burnout. Eight items are reverse scored.
Mean Change from Baseline in Teacher Burnout Scores on the Maslach Burnout Inventory at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher self-report with a 23-item scale (Maslach & Jackson, 1981) measured on a 7-point Likert scale, where 1=Never, 2=A few times, 3=Once a month or less, 4=A few times a month, 5=Once a week, 6=A few times a week, 7=Every day. Mean score calculated, with higher scores indicating higher levels of burnout. Eight items are reverse scored.

SECONDARY OUTCOMES:
Mean Change from Baseline in Student Anxiety Scores on the Anxiety Subscale of the Seattle Personality Questionnaire at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Student self-report with a 7-item scale (Kusche et al., 1988; Rains, 2003) measured on a 4-point Likert scale, where 1=Not at all, 2=A little bit, 3=Sometimes, 4=Always. Mean score calculated, with higher scores indicating higher levels of anxiety. No reverse scored items.
Mean Change from Baseline in Student Anxiety Scores on the Anxiety Subscale of the Seattle Personality Questionnaire at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Student self-report with a 7-item scale (Kusche et al., 1988; Rains, 2003) measured on a 4-point Likert scale, where 1=Not at all, 2=A little bit, 3=Sometimes, 4=Always. Mean score calculated, with higher scores indicating higher levels of anxiety. No reverse scored items.
Mean Change from Baseline in Classroom Supportiveness Scores on the Classroom Supportiveness Subscale of the Sense of Classroom as a Community Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Student self-report with a 14-item scale (Battistich et al., 1995; 1997) measured on a 5-point Likert scale, 1=Disagree a lot, 2=Disagree a little, 3=Don't agree or disagree, 4=Agree a little, 5=Agree a lot. Mean score calculated, with higher scores indicating higher levels of classroom supportiveness. Three items are reverse scored.
Mean Change from Baseline in Classroom Supportiveness Scores on the Classroom Supportiveness Subscale of the Sense of Classroom as a Community Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Student self-report with a 14-item scale (Battistich et al., 1995; 1997) measured on a 5-point Likert scale, 1=Disagree a lot, 2=Disagree a little, 3=Don't agree or disagree, 4=Agree a little, 5=Agree a lot. Mean score calculated, with higher scores indicating higher levels of classroom supportiveness. Three items are reverse scored.
Mean Change from Baseline in Teacher General Teaching Efficacy Scores on the General Teaching Efficacy Scale on the Teacher Efficacy Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher self-report with a 10-item scale (Woolfolk et al., 1990) measured on a 5-point Likert scale, where 1=Strongly Disagree, 2=Disagree, 3=Unsure, 4=Agree, 5=Strongly Agree. Mean score calculated, with higher scores indicating higher levels of general teaching efficacy. Six items are reverse scored.
Mean Change from Baseline in Teacher General Teaching Efficacy Scores on the General Teaching Efficacy Scale on the Teacher Efficacy Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher self-report with a 10-item scale (Woolfolk et al., 1990) measured on a 5-point Likert scale, where 1=Strongly Disagree, 2=Disagree, 3=Unsure, 4=Agree, 5=Strongly Agree. Mean score calculated, with higher scores indicating higher levels of general teaching efficacy. Six items are reverse scored.
Mean Change from Baseline in Teacher Self-Awareness Scores on the Self-Awareness Scale at 14 weeks and 6-month follow-up | From baseline to end of intervention at 14 weeks
  Teacher self-report with a 6-item scale (American Institutes for Research & Collaborative for Academic, Social, and Emotional Learning, 2013) measured on a 4-point Likert scale, 1=Rarely, 2=Occasionally, 3=Frequently, 4=Almost Always. Mean score calculated, with higher scores indicating higher levels of self-awareness. No reverse scored items.
Mean Change from Baseline in Teacher Self-Awareness Scores on the Self-Awareness Scale at 14 weeks and 6-month follow-up | From 14 weeks to 6 months after the end of intervention
  Teacher self-report with a 6-item scale (American Institutes for Research & Collaborative for Academic, Social, and Emotional Learning, 2013) measured on a 4-point Likert scale, 1=Rarely, 2=Occasionally, 3=Frequently, 4=Almost Always. Mean score calculated, with higher scores indicating higher levels of self-awareness. No reverse scored items.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Schonert-Reichl, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD)(de-identified) will be made available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD and any additional supporting information will become available starting 6 months after publication and will be available for 5 years afterwards.
Access Criteria: Requests for IPD can be made in writing to the Study Principal Investigator, for all types of analyses and via all mechanisms. Release of IPD is contingent upon receipt of Institutional Review Board (IRB) approval documentation or other determination.

REFERENCES:
- [Background] Schonert-Reichl KA. Relations of peer acceptance, friendship adjustment, and social behavior to moral reasoning during early adolescence. The Journal of Early Adolescence. 1999; 19(2): 249-279.
- [Background] Wentzel KR, Barry CM, Caldwell KA. Friendships in middle school: Influences on motivation and school adjustment. Journal of Educational Psychology. 2004. 96: 195-203. http://dx.doi.org/10.1037/\0022-0663.96.2.195
- [Background] Oberle E, Schonert-Reichl KA, Thomson KC. Understanding the link between social and emotional well-being and peer relations in early adolescence: gender-specific predictors of peer acceptance. J Youth Adolesc. 2010 Nov;39(11):1330-42. doi: 10.1007/s10964-009-9486-9. Epub 2009 Nov 29. PMID 20091211
- [Background] Noam GG, Goldstein LS. The Resilience Inventory. 1994. Unpublished protocol.
- [Background] Song M. Two studies on the resilience inventory (RI): Toward the goal of creating a culturally sensitive measure of adolescent resilience. Dissertation Abstracts International. 2003. 64 (8B). (UMI No. 3100166) Harvard: ProQuest Information and Learning
- [Background] Kusche CA, Greenberg MT, Beilke R. Seattle Personality Questionnaire for young school-aged children. Unpublished manuscript. 1988. University of Washington, Department of Psychology, Seattle.
- [Background] Rains C. Seattle Personality Questionnaire-Original (Fast Track ProjectTechnical Report). 2003. Retrieved October 2005 from sanford.duke.edu/centers/child/fasttrack/techrept/s/spq/spq3tech.pdf
- [Background] Kam C, Greenberg MT. Technical measurement report on the teacher social competence rating scale. Unpublished technical report. 1998. Prevention Research Center for the Promotion of Human Development, The Pennsylvania State University
- [Background] Battistich V, Solomon D, Watson M, Schaps E. Caring school communities. Educational Psychologist. 1997. 32: 137 - 151.
- [Background] Neff KD. The development and validation of a scale to measure self-compassion, Self and Identity. 2003. 2: 223-250.
- [Background] Roeser RW, Schonert-Reichl KA, Jha A, Cullen M, Wallace L, Wilensky R, Oberle E, Thomson K, Taylor C, Harrison J. Mindfulness training and reductions in teacher stress and burnout: Results from two randomized, waitlist-control field trials. Journal of Educational Psychology. 2013. 105(3): 787-804.
- [Background] Pettegrew LS, Wolf GE. Validating measures of teacher stress. American Educational Research Journal. 1982. 19(3): 373-396.
- [Background] Maslach C, Jackson SE. The measurement of experienced burnout. Journal of Occupational Behaviour. 1981. 2: 99-113.
- [Background] Woolfolk AE, Rosoff B, Hoy WK. Teachers' sense of efficacy and their beliefs about managing students. Teaching and Teacher Education. 1990. 6: 137-148.
- [Background] American Institutes for Research and Collaborative for Academic, Social, and Emotional Learning. Student self-report of social and emotional competencies. 2013. Washington DC and Chicago: Authors.
- [Background] Bandura A, Barbaranelli C, Caprara GV, Pastorelli C. Mechanisms of moral disengagement in the exercise of moral agency. Journal of Personality and Social Psychology. 1996. 71: 364-374.
- [Background] Parkhurst JT, Asher SR. Peer rejection in middle school: Subgroup differences in behavior, loneliness, and interpersonal concerns. 1992. Developmental Psychology. 28(2): 231-241. Doi:10.1037/0012-1649.28.2.231
- [Background] Battistich V, Solomon D, Watson M, Schaps E. Schools as communities, poverty levels of student populations, and students' attitudes, motives, and performance: A multilevel analysis. 1995. American Educational Research Journal. 32: 627-658.
- [Background] Miller R. Tales of teacher absence: New research yields patterns that speak to policymakers. 2008. Center for American Progress: Washington, DC.
- [Background] Colaianne BA, Galla BM, Roeser RW. Perceptions of mindful teaching are associated with longitudinal change in adolescents' mindfulness and compassion. 2020. International Journal of Behavioral Development. 44(1): 41-50.
- [Background] Harris AR, Jennings PA, Katz DA, Abenavoli RM, Greenberg MT. Promoting stress management and wellbeing in educators: Feasibility and efficacy of a school-based yoga and mindfulness intervention. 2015. Mindfulness. 7(1): 143-154. http://dx.doi.org/10.1007/s12671-015-0451-2.
- [Background] Jennings PA, Brown JL, Frank JL, Doyle S, Oh Y, Davis R, Rasheed D, DeWeese A, DeMauro AA, Cham H, Greenberg MT.Impacts of the CARE for Teachers Program on teachers' social and emotional competence and classroom interactions. 2017. Journal of Educational Psychology. 109(7): 1010-1028. https://doi.org/10.1037/edu0000187
- [Background] Kemeny ME, Foltz C, Cavanagh JF, Cullen M, Giese-Davis J, Jennings P, Rosenberg EL, Gillath O, Shaver PR, Wallace BA, Ekman P. Contemplative/emotion training reduces negative emotional behavior and promotes prosocial responses. Emotion. 2012 Apr;12(2):338-50. doi: 10.1037/a0026118. Epub 2011 Dec 12. PMID 22148989
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Merikangas KR, Walters EE. Lifetime prevalence and age-of-onset distributions of DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):593-602. doi: 10.1001/archpsyc.62.6.593. PMID 15939837
- [Background] Lever N, Mathis E, Mayworm A. School Mental Health Is Not Just for Students: Why Teacher and School Staff Wellness Matters. Rep Emot Behav Disord Youth. 2017 Winter;17(1):6-12. No abstract available. PMID 30705611
- [Background] Lomas T, Medina JC, Ivtzan I, Rupprecht S, Eiroa-Orosa FJ. The impact of mindfulness on the wellbeing and performance of educators: A systematic review of the empirical literature. 2017. Teaching and Teacher Education. 61: 132-141. https://doi.org/10.1002/sop2.16
- [Background] Merikangas KR, Nakamura EF, Kessler RC. Epidemiology of mental disorders in children and adolescents. Dialogues Clin Neurosci. 2009;11(1):7-20. doi: 10.31887/DCNS.2009.11.1/krmerikangas. PMID 19432384
- [Background] Roeser RW, Galla BM, Baelen RN. Evidence on the impacts of school-based mindfulness programs on student outcomes in P-12 educational settings [Issue Brief]. 2020. Edna Bennett Pierce Prevention Research Center. https://www.prevention.psu.edu/uploads/files/RWJF-Mindfulness-Brief-Dec2020.pdf
- [Background] Schonert-Reichl KA. Social and emotional learning and teachers. 2017. Future of Children. 27: 137-155.
- [Background] Schonert-Reichl KA, Lawlor MS. The effects of a mindfulness-based education program on pre-and early adolescent's well-being and social and emotional competence. 2010. Mindfulness. 1 (1): 137-151.
- [Background] Schonert-Reichl KA, Oberle E, Lawlor MS, Abbott D, Thomson K, Oberlander TF, Diamond A. Enhancing cognitive and social-emotional development through a simple-to-administer mindfulness-based school program for elementary school children: a randomized controlled trial. Dev Psychol. 2015 Jan;51(1):52-66. doi: 10.1037/a0038454. PMID 25546595
- [Background] Theokas C, Lerner RM. Observed ecological assets in families, schools, and neighborhoods: Conceptualization, measurement, and relations with positive and negative developmental outcomes. 2006. Applied Developmental Science. 10: 61-74.